CLINICAL TRIAL: NCT03395249
Title: A Two-part, Double-blind, Placebo-controlled, Phase I Study of the Safety, Tolerability and Pharmacokinetics of SPR994 Following Single and Multiple Ascending Doses of SPR994 Administered Orally in Healthy Volunteers
Brief Title: Phase 1 Study of Safety, Tolerability and Pharmacokinetics of SPR994
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: CPR Pharma Services Pty Ltd, Australia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPR994-101
Record Dates: First submitted 2017-10-19; First posted 2018-01-10 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
Keywords: safety; tolerability; pharmacokinetics; SPR994
MeSH Terms: interventions — tebipenem

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects will be randomized in a 3:1 ratio of SPR994 to placebo. Study drug tablets, both active and placebo, are the same shape, weight and size. Those blinded to study drug assignment include the sponsor, the PI, clinical study personnel participating in subjects' care or clinical evaluations, and the subjects. Those unblinded to study drug assignment include the statisticians preparing the randomisation, pharmacy personnel, the unblinded study monitor, the bioanalytical laboratory, and the pharmacokineticist performing interim PK analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPR994, FI, F2, F3, F4 Oral Tablets (Experimental): SPR994 is active against multidrug-resistant Gram-negative and Gram-positive pathogens that cause serious and life-threatening infections, including extended spectrum beta-lactamase (ESBL) producers as well as strains resistant to levofloxacin and trimethoprim/sulfamethoxazole. SPR994 is administered in tablet form orally. Up to five different time released formulations of SPR994 will be studied in this protocol at 100 mg, 300 mg, 600 mg and 900 mg dosages.
  SAD Cohorts: One dose (two for food effect cohort) MAD Cohorts: Twenty-seven (27) doses administered twice daily (BID) over a period of 14 days or forty doses administered three times daily (TID) over period of 14 days
  Interventions: Drug: SPR994
- Placebo Oral Tablet (Placebo Comparator): Placebo tablets (100, 300, and 600 mg) are pressed from a single placebo blend consisting of the same inactive ingredients; the active pharmaceutical ingredient (API) is replaced by Mannitol 200SD.
  SAD Cohorts: One dose (two for food effect cohort) MAD Cohorts: Twenty-seven (27) doses administered BID over a period of 14 days or forty doses administered TID over a period of 14 days
  Interventions: Drug: Placebo Oral Tablet
- Optional Orapenem Open-Label Control (Other): A single, optional, open-label, control cohort that may enroll, in which all 8 subjects receive Orapenem.
  SAD Cohort: One dose under fasted conditions and one dose under fed conditions.
  Interventions: Drug: Orapenem®

INTERVENTIONS:
Drug: SPR994 — SAD: Double-blind dosing will occur in all SAD Cohorts except for Cohort 12. In each cohort, six subjects will receive one of five different timed release formulations of SPR994 and 2 subjects will receive placebo. Subjects in SAD Cohorts 2, 3, 6, 16 and 17 will receive a single dose following a 10-h fast. Subjects in SAD Cohorts 1, 8-15 will receive one dose of SPR994 or placebo following a 10-h fast on Day 1 and a second dose following consumption of a standardized meal on Day 7. The dose escalation steps may be altered following review of the safety data of each cohort.
  MAD: Double-blind dosing will occur in all MAD Cohorts. Subjects will receive multiple doses of an optimal timed release formulation of SPR994 in MAD Cohort 4 (300 mg) and Cohort 5 (600 mg) or placebo for 14 consecutive days at either BID or TID dosing beginning on Day 1.
  Other Names: SPR994 Oral Tablet
  Arms: SPR994, FI, F2, F3, F4 Oral Tablets
Drug: Placebo Oral Tablet — Mannitol 200SD SAD: Two subjects in each cohort will receive matching placebo. MAD: Two participants in each cohort will receive matching placebo.
  Other Names: Placebo
  Arms: Placebo Oral Tablet
Drug: Orapenem® — Tebipenem pivoxil granules
  Other Names: Orapenem® fine granules
  Arms: Optional Orapenem Open-Label Control

SUMMARY:
This is a double-blind, placebo-controlled, ascending dose, multi-cohort trial. The study will be conducted in 2 parts: a single ascending dose (SAD) part, followed by a multiple ascending dose (MAD) part. In SAD, all subjects will receive 1 dose of SPR994 (100, 300, 600 or 900 mg) or placebo, except for subjects enrolled in food effect cohorts in which subjects will receive one dose following a 10 hour fast and a second dose in the fed state following a minimum 5 days washout period. There is a single, optional, open-label control cohort that may enroll, in which all 8 subjects will receive Orapenem® (tebipenem pivoxil fine granules). In MAD, subjects will receive multiple doses of SPR994 (300 or 600 mg) or placebo for 14 consecutive days at either BID or TID dosing. In both parts, cohorts will be exposed to increasing doses of SPR994 with various extended release formulations.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial. Up to one hundred fifty two (152) subjects aged 18-55, who fulfill the inclusion/exclusion criteria, may be enrolled in this study. Up to a total of 17 SAD and 2 MAD cohorts of eight subjects each will be examined. Subjects in each cohort will be randomized 3:1 to receive SPR994 at doses ranging from 100 mg to 900 mg or placebo in various immediate and timed release formulations. One SAD control cohort, Cohort 12, may be enrolled in which eight subjects will receive a single dose of Orapenem® at 300 mg in a fed and fasted state. Dosing is complete in SAD Cohorts 1-3, 6 and 7. Subjects in Cohorts 1-3 received a single dose of SPR994 and subjects in food effect Cohorts 6 and 7 each received 2 doses. Subjects enrolled in SAD Cohorts 8 and beyond will receive a single dose of SPR994 or placebo in a fasted state and a second dose following a standardized meal to investigate food effect on the pharmacokinetics of SPR994 and TBPM. SAD Cohorts 8 through 10 may run in a staggered or concurrent manner before enrollment of further cohorts. Blinded pharmacokinetic data will be reviewed at the conclusion of Cohort 10 (300 mg fasted & fed). Should the PK be optimized in one of the various time released formulations, the Sponsor may decide to proceed to enrollment of the 600 mg Cohorts using the optimal formulation; other timed release formulations may also be explored at 300 mg dose in a staggered or concurrent manner until an optimal formulation(s) is identified. When an optimal formulation(s) is identified, the 600 mg Cohorts may run in a staggered or concurrent manner. SAD Cohorts 16 (100 mg fasted) and 17 (900 mg fasted) may run prior to or in a staggered or concurrent manner with MAD Cohorts 4 (300 mg) and 5 (600 mg). During the MAD part of the study, subjects will receive 27 doses of SPR994 or placebo over a period of 14 days. Based on the observed PK of SPR994 in prior cohorts, the total number of doses may be increased to 40 doses of SPR994 or placebo administered TID over 14 days; only one dose will be administered on Day 14 to allow for PK sample collection In both SAD and MAD parts of the study, the Cohorts will be exposed to increasing doses of SPR994. Each part (SAD and MAD) of the study will consist of 3 periods: a screening period, a treatment period, and a follow-up period. The safety and tolerability of SPR994 will be assessed based on the types and frequency of adverse events (AEs) reported; concomitant medication usage; and changes from baseline in physical examination, weight, vital signs, ECG, and standard clinical laboratory tests. A Safety Management Group (SMG) will review the data of cohorts prior to escalating to the next dose level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males and/or females (of non-childbearing potential), 18 to 55 years of age (inclusive) at the time of screening;
* Body mass index ≥ 18.5 and ≤ 29.9 (kg/m2) and 55.0 and 100.0 kg (inclusive) for all cohorts;
* Medically healthy without clinically significant (CS) abnormalities at the screening visit or Day -1, including:

  1. Physical examination, vital signs including temperature, heart rate, respiratory rate, and blood pressure;
  2. Triplicate electrocardiograms (ECGs) taken at least 1 minute apart with QT wave corrected for heart rate (HR) using Fridericia's method (QTcF) interval duration less than 450 msec obtained as an average from the triplicate screening and pre-dose Day 1 ECGs after at least 5 min in a semi-supine quiet rest;
  3. Haemoglobin > 12.5, haematocrit 37%, white blood cell (WBC) count > 3.5, or platelet count equal to or greater than the lower limit of normal range of the reference laboratory (may be confirmed upon repeat analysis);
  4. Creatinine, blood urea nitrogen (BUN), equal to or less than the upper limit of normal; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) equal to or < 1.5 times the upper limit of normal for the reference laboratory and confirmed on repeat analysis; results of all other clinical chemistry and urine analytes without any CS abnormality.

Discussion between the PI and the Sponsor Medical Monitor is encouraged regarding any abnormal laboratory value that is outside of the normal range during the pre-dose period.

* Be non-smokers (including tobacco, e-cigarettes or marijuana) for at least 1 month prior to participation in the study;
* Willing and able to provide written informed consent;
* Be willing and able to comply with all study assessments and adhere to the protocol schedule;
* Have suitable venous access for blood sampling;
* If female, be of non-childbearing potential (e.g. post-menopausal as demonstrated by follicle stimulating hormone or surgical sterilization i.e., tubal ligation or hysterectomy). Provision of documentation is not required for female sterilization, verbal confirmation is adequate;
* If male, a willingness not to donate sperm and if engaging in sexual intercourse with a female partner who could become pregnant, a willingness to use a condom in addition to having the female partner use a highly effective method of birth control (such as an intrauterine device, diaphragm, oral contraceptives, injectable progesterone, subdermal implants, or a tubal ligation). This criterion applies to males (and/or female partners) who are surgically sterile and must be followed from the time of first study drug administration until 30 days after the final administration of study drug.

Exclusion Criteria:

* History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or surgery within the past 3 months determined by the PI to be clinically relevant;
* History of known or suspected Clostridium difficile infection;
* History of seizure disorders, except for a single febrile seizure in childhood;
* Positive urine drug/alcohol testing at screening or Day -1;
* Positive testing for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibodies (HCV);
* History of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where 1 standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years;
* Use of any prescription medication or any over-the-counter medication, including herbal products and vitamins within 7 days prior to randomization;
* Documented hypersensitivity reaction or anaphylaxis to any medication;
* Donation of blood or plasma within 30 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrollment;
* Participation in another investigational clinical trial within 30 days prior to Day 1;
* Any other condition or prior therapy, which, in the opinion of the PI, would make the volunteer unsuitable for this study, including unable to cooperate fully with the requirements of the study protocol or likely to be non-compliant with any study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Safety measures: adverse events | SAD: 1 to 7 days or 1 to 13 (food effect cohort); MAD 1 to 20 days
  The incidence and severity of AEs
Safety measures: concomitant medications | SAD: 1 to 7 days or 1 to 13 (food effect cohort); MAD: 1 to 20 days
  The type and frequency of medications used
Safety measures: physical examination | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: weight | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: pulse rate | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: ECG | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: clinical laboratory testing | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: respiratory rate | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: blood pressure | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit
Safety measures: body temperature | SAD: -1 to 7 days or -1 to 13 (food effect cohort); MAD: -1 to 20 days
  Change from baseline to end of study visit

SECONDARY OUTCOMES:
Pharmacokinetics: Time to maximum concentration (Tmax) | SAD: Day 1 to Day 3 and Day 7 to 9 (Food Effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Maximum concentration (Cmax) | SAD: Day 1 to Day 3 and Day 7 to 9 (Food Effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Area under the concentration-time curve from time 0 to last measurable time-point (AUC0-t) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Area under the concentration-time curve from time 0 to infinity (AUC0-inf) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Terminal Elimination Rate Constant (kel) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Terminal half-life (t1/2) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Terminal clearance (CL/F) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Volume of distribution | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: Area under the concentration-time curve from 0 to 12 hours from the start of first dose (AUC0-12h) | SAD: Day 1 to Day 3 and Day 7 to 9 (food effect); MAD Day 1 to 16
  Plasma Sample Collection for PK Analysis:
  SAD Cohorts 1 and 7: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 2, 3, and 6: Day 1 at the same time-points as SAD Cohorts 1 and 7. SAD Cohorts 8 - 15: Days 1 and 7 (Food Effect Cohorts) at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12, 24, and 48 h post-dose.
  SAD Cohorts 16 and 17: Day 1 at the same time-points as SAD Cohorts 8 - 15. MAD Cohorts 4 and 5: Day 1 at pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8, 12 h following start of the first dose (BID dosing) or pre-dose and at 15, 30, 45 min and 1, 1.5, 2, 4, 6 and 8 h following start of first dose and prior to second dose (TID dosing); Prior to the morning dose on Days 2, 3, 5, 7, 9, 11 and 13; Pre-dose, 15, 30, 45 min and 1, 1.5, 2, 4, 6, 8
Pharmacokinetics: SPR994 excreted in urine in each collection interval | SAD: Days 1-2 and 7-8 (food effect cohorts). MAD: Day 1-2 and 14-15.
  SAD: Urine samples for PK will be collected at pre-dose and during the following intervals(total collection): 0-4, 4-8, 8-12, and 12-24 hours after dosing.
  MAD: Urine samples for PK will be collected at pre-dose on Day 1 and during the followingintervals (total collection): 0-4, 4-8, and 8-12 hours after start of first dose (BID dosing) or pre-dose on Day 1 and during the following intervals (total collection): 0-4, 4-8 prior to next dose (Days 1-2); and 0-4, 4-8, 8-12, and 12-24 hours following start of the last dose (Days 14-15).

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Lemech, FRACP, MD, Principal Investigator — Scientia Clinical Research Limited
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

REFERENCES:
- [Derived] Eckburg PB, Jain A, Walpole S, Moore G, Utley L, Manyak E, Dane A, Melnick D. Safety, Pharmacokinetics, and Food Effect of Tebipenem Pivoxil Hydrobromide after Single and Multiple Ascending Oral Doses in Healthy Adult Subjects. Antimicrob Agents Chemother. 2019 Aug 23;63(9):e00618-19. doi: 10.1128/AAC.00618-19. Print 2019 Sep. PMID 31262768